CLINICAL TRIAL: NCT06247579
Title: Effects of Dietary Polystyrene Microplastics From Disposable Plastic Tableware on Anxiety- and Depression-like Behaviors
Brief Title: Effects of Dietary Polystyrene Microplastics on Anxiety- and Depression-like Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, WenJing Zhao, M.D.; attending doctor, Northern Jiangsu People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Dietary
Record Dates: First submitted 2024-01-07; First posted 2024-02-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Depression, Anxiety
Keywords: Gut microbiome; Anxiety; Depression; Polystyrene microplastics
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The exposure group will use disposable plastic tableware (DPT) made of polystyrene, provided by the hospital canteens for two months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): The control group, consisting of resident physicians, will use non-disposable plastic tableware (NDPT) provided by hospital canteens for two months.
- The exposure group (Experimental): The exposure group, also comprising resident physicians, will use disposable plastic tableware (DPT) made of polystyrene, provided by the same hospital canteens for two months
  Interventions: Other: Dietary polystyrene microplastics from disposable plastic tableware

INTERVENTIONS:
Other: Dietary polystyrene microplastics from disposable plastic tableware — Microplastic release from the daily use of disposable plastic materials (e.g., plastic boxes) when holding hot food or drink.
  Arms: The exposure group

SUMMARY:
The objective of this clinical trial is to explore the potential impact of dietary polystyrene microplastics on anxiety- and depression-like behaviors in resident physicians. Specifically, the study aims to address two key questions:

1. Can dietary polystyrene microplastics induce alterations in the human gut microbiome?
2. Can dietary polystyrene microplastics exacerbate anxiety- and depression-like behaviors?

Participants will be divided into two groups based on their habitual eating practices: The control group, consisting of resident physicians, will use non-disposable plastic tableware (NDPT) provided by hospital canteens for two months. In contrast, the exposure group, also comprising resident physicians, will use disposable plastic tableware (DPT) made of polystyrene, provided by the same hospital canteens, over the same period.

DETAILED DESCRIPTION:
The mental health and well-being of resident physicians is a critical topic that has gained increasing attention recently. Recent studies have shown a growing prevalence of mental health illnesses worldwide. For medical trainees and resident physicians, high rates of depression, anxiety, suicidal ideation, and burnout have been consistently observed. Moreover, contemporary research suggests that dietary exposure plays a pivotal role in the development of mental illnesses. Disposable plastic tableware, commonly used during resident training programs, could be a contributing factor. However, the specific effects of dietary exposure from such tableware on mental health, particularly through the gut-brain axis, remain largely unexplored. Consequently, investigating the potential impact of dietary polystyrene microplastics on anxiety- and depression-like behaviors in resident physicians is essential.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer resident physician at the base of Northern Jiangsu Hospital, Yangzhou, China

Exclusion Criteria:

* received chemotherapy, radiotherapy, or surgery in the 3 -6 months before sampling
* diagnosed with mental illness
* diagnosed with digestive system diseases

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Assessing mental status using the depression anxiety stress scales-21 (DASS-21) questionnaire | At the baseline and end of this clinical trial an average of two months. the enrolled participants will be asked to complete the DASS-21 questionnaire.
  In this study, the researchers utilized the Chinese version of the Depression Anxiety Stress Scales-21 (DASS-21), a widely recognized and reliable instrument for assessing depression, anxiety, and stress. This comprehensive tool is divided into three sections, each dedicated to evaluating the levels of depression, anxiety, and stress, respectively. The depression scale scores range from 0 to 21, with normal scores falling below 4. Anxiety scores also range from 0 to 21, with normal scores below 3. For stress, scores range from 0 to 18, with scores below 7 considered normal. Higher scores on any of these scales indicate elevated levels of depression, anxiety, or stress. In this research, the DASS-21 was employed to monitor the variations in anxiety and depression-like behaviors among the two groups, both at baseline and after the treatment period.

SECONDARY OUTCOMES:
Alterations in human gut microbial diversity investigated through 16S rRNA | At the beginning and conclusion of this clinical trial, spanning an average duration of two months, the enrolled participants will be asked to provide fecal samples
  The gut microbiota encompasses the microorganisms residing in the human gastrointestinal tract. Microbial diversity refers to the variety of different species present in the gut microbiome. In this study, DNA extraction from fecal samples is carried out in two primary steps. Initially, the sample undergoes purification using multiple reagents and centrifugation. This process isolates the microbes by removing other fecal components. The next step involves lysing bacterial cells; this is achieved by incubating the samples in lysis buffer with agitation. Subsequently, the extracted DNA is amplified through techniques such as multiple displacement amplification. A 16S rRNA primer is then selected for gene sequencing. The sequences obtained from the 16S rRNA will be analyzed to ascertain the gut microbial diversity at the species level.

CONTACTS AND LOCATIONS:
Locations (1):
- Ju Gao, Yangzhou, Jiangsu, China